CLINICAL TRIAL: NCT01640639
Title: Effects of Thalidomide on Left Ventricular Morphology and Function in Patients With Congestive Heart Failure - The THUNDER Trial
Brief Title: THalidomide on Left ventricUlar Morphology aND Function in congEstive heaRt Failure
Acronym: THUNDER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 430/2012/D
Record Dates: First submitted 2012-07-06; First posted 2012-07-16 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Congestive Heart Failure
Keywords: left ventricular function
MeSH Terms: conditions — Heart Failure | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide (Active Comparator): Thalidomide
  Interventions: Drug: Thalidomide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — Thalidomide, pill, 50 mg, once p.d., 6 weeks
  Arms: Thalidomide
Drug: Placebo — Placebo, pill, once p.d., 6 weeks
  Arms: Placebo

SUMMARY:
Several studies have shown that inflammation and matrix degradation have pathogenic effects on the myocardium by influencing heart contractility, inducing hypertrophy, degrading the matrix, or enhancing fibrosis, thus contributing to the continuous myocardial remodeling process.

The sedative and antinausea drug thalidomide has been shown to have both anti-inflammatory and antioncogenic properties that could be of benefit in case of congestive heart failure (CHF).

Previous, small investigations have shown an improvement in left ventricular ejection fraction and a favorable cardiac remodeling during thalidomide therapy.

DETAILED DESCRIPTION:
Purpose

Several studies have shown that inflammation and matrix degradation have pathogenic effects on the myocardium by influencing heart contractility, inducing hypertrophy, degrading the matrix, or enhancing fibrosis, thus contributing to the continuous myocardial remodeling process.

The sedative and antinausea drug thalidomide has been shown to have both anti-inflammatory and antioncogenic properties that could be of benefit in case of congestive heart failure (CHF).

Previous, small investigations have shown an improvement in left ventricular ejection fraction and a favorable cardiac remodeling during thalidomide therapy.

Purpose

The primary objective of this study is to carry out a double-blind, randomized, placebo-controlled study to assess the effects of oral thalidomide on left ventricular morphology and function in patients with CHF

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction < 50%
* Signs and symptoms of stable CHF
* NYHA III or IV functional class

Exclusion Criteria:

* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT
* Clinical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction | baseline and 6 months
  changes in left ventricular ejection fraction at 6 months as compared with baseline

SECONDARY OUTCOMES:
Changes in NYHA functional class | baseline and 6 months
  changes in NYHA functional class at 6 months as compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University La Sapienza, Rome, Italy